CLINICAL TRIAL: NCT01705821
Title: Measuring Forces Applied During Skull Base Surgery
Brief Title: Forces During Skull Base Surgery
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Robert Webster, Assistant Professor, Vanderbilt University
Other Study IDs: 121194
Record Dates: First submitted 2012-10-08; First posted 2012-10-12 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2014-12

CONDITIONS: Skull Base; Pituitary; Robotics; Endonasal Surgery; Sinus Surgery
Keywords: Skull base; Pituitary; Robotics; Endonasal surgery; Sinus surgery
MeSH Terms: conditions — Pituitary Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Skull Base Surgery Candidate: Patient with a skull base lesion will undergo use of standard surgical curette with force sensor built into shaft. 6-axis force and torque data will be collected during the surgical procedure.
  Interventions: Device: Use of force sensing surgical curette; Procedure: Removal of pituitary tumor using modified curette

INTERVENTIONS:
Device: Use of force sensing surgical curette — Use of a standard surgical curette outfitted with an in-line 6-axis force and torque transducer for collection of force data during surgery.
Procedure: Removal of pituitary tumor using modified curette

SUMMARY:
This study is designed to measure forces applied using standard surgical instruments at the skull base during resection of skull base lesions. This data will be useful for optimizing an active canula robot for assisting in skull base surgery. We hypothesize that through measurement of forces generated during routine endoscopic skull base surgery we will be able to optimize the canulas of an active canula robot for skull base surgery.

DETAILED DESCRIPTION:
At some time in their lives, 1 in 5 people will have a pituitary tumor, and 1 in 600 of these will have the tumor grow large enough (>1 cm in diameter) that surgical resection is required. Traditionally, surgery to remove pituitary tumors or other tumors at the skull base requires transcranial or transfacial access. In these approaches, large traumatic, often disfiguring, openings must be created in the patient's forehead or cheek. Endonasal skull base surgery reduces invasiveness resulting in less trauma, fewer complications, and shorter surgical time. However, despite the compelling advantages for the patient, only a small percentage of skull base surgeries are done endonasally. While exact statistics are not available, the current best estimate in the literature is that less than 50% and most likely less than 20% of these tumors are addressed by endonasal surgery.

The endonasal approach is underemployed despite its demonstrated benefits to the patient because existing surgical instruments have limited dexterity and approach angles, and simultaneously manipulating several of them through a nostril while performing complex surgical procedures is so technically challenging that only a small number of expert surgeons can accomplish it. Even for these experts, mortality rates are non-negligible (0.9%), and there remain contraindications to the endonasal approach, including occlusion of the surgical site by delicate and critical neurovascular structures (e.g. carotid arteries, optic nerves), inability to fully reconstruct the dura due to lack of surgical tool dexterity, and long surgical duration. All of these contraindications are directly related to limitations in instrument dexterity and visualization, which motivates the development of a robotic system for endonasal skull base surgery. Such a robot can potentially increase surgical dexterity and reduce the technical complexity of the procedure for surgeons, thereby increasing the percentage of patient who benefit from the endonasal technique.

While many robotic systems have been developed for intravascular interventions as well as natural orifice surgery though other orifices, comparatively few systems have been targeted at endonasal surgery. This is likely due to the smaller size of the nasal cavity and nostril compared to other natural orifices.

For endonasal robots, the limited space available in the nostril opening, combined with the need to work dexterously within the cavities in the head, implies that instrument shafts must be small in diameter while enabling dexterous motions of instrument tips. A recently invented robot design that matches these characteristics is the concentric tube robot concept, which is also known as by the name active cannula.

A robot suitable for endonasal surgery is being developed (see reference #3), however in order to optimize this robotic system, intraoperative data must be obtained to determine how the robot interacts with the patient's tissues. The aim of this study is to modify a traditional tool used in the operating room to allow determination of forces at the skull base on both hard and soft tissues. This surgical curette will be used in the standard fashion during endonasal skull base surgery, however will provide valuable information.

The modified curette will consist of two segments joined by a Nano17 6-axis force sensor. (Image 1) The force sensor is integrated into the shaft of the instrument (a standard neurosurgical ring curette) and insulated from the shaft with two polyetherimide (also known as ULTEM) disks so that no current can be transmitted from the force sensor to the curette. The sensor is held to the shaft by medical grade adhesive and set screws.

The patients will be recruited from the PIs clinical practice. Informed consent will be obtained. At the appropriate time during surgery this curette will be used to collect force date. This force transducer operates at 5V (4.8-9V range). These transducers are commonly used in medical and dental research (see reference #5).

No additional operating room or anesthesia time will be required.

ELIGIBILITY:
Inclusion criteria:

* Any male or female patient 18-75 years old undergoing endonasal skull base surgery for a skull base lesion.
* Competent in decision making process and able to sign a written informed consent form.

Exclusion Criteria:

-Any patient not able to give written informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients undergoing standard endonasal skull base surgery.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2012-10; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
6-axis force and torque data from routine endoscopic transnasal skull base surgery | 12 months
  This data will be collected and recorded via a computer interface with our sensorized tool and recorded in standard units for force and torque. We will also look at the variability of forces between patients after collecting this data. The data will be useful in optimizing a robotic system for endonasal surgery as described in the secondary outcome measure.

SECONDARY OUTCOMES:
Percent tumor removal in skull and cadaver studies | 12 months
  The force and torque data will allow our team of Engineers to optimize our robotic system to be best suited for removing pituitary tumors transnasally. The robot consists of specially designed flexible arms with end effectors that each need to be able to withstand and produce the necessary forces to complete pituitary tumor excision. This will be measured by optimizing our robot based on the findings in the primary outcome measure and then evaluating the robot for efficiency and effectiveness of mock pituitary tumor removal from skull and cadaver specimens. We will investigate percent tumor removal and speed of tumor removal once the robot is optimized.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Webster, PhD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Skull Base Center, Nashville, Tennessee, United States